CLINICAL TRIAL: NCT04179032
Title: A Multi-Center, Open-Label Trial to Evaluate the Pharmacokinetics, Safety, and Pharmacodynamics of Subcutaneously Administered Belimumab, a Human Monoclonal Anti-BLyS Antibody, Plus Standard Therapy in Pediatric Participants With Systemic Lupus Erythematosus (SLE)
Brief Title: Study of Subcutaneous (SC) Belimumab in Pediatric Participants With Systemic Lupus Erythematosus (SLE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200908; 2023-509413-37-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; Pediatric; Pharmacokinetics; Pharmacodynamics; Safety; Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: Cohorts 1, 2, and 3 will be recruited in parallel design. In Part A participants will receive 200 mg/mL belimumab via SC injection once a week (QW) in Cohort 1, every 10 days (Q10d) in Cohort 2, and every 2 weeks (Q2W) in Cohort 3. In Part B, dosing frequency may change according to pre-defined criteria based on changes in body weight of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belimumab 200 mg (Experimental): Participants with Systemic Lupus Erythematosus were administered with Belimumab 200 milligram per milliliter (mg/mL) subcutaneous (SC) injection. The dosing frequency was based on body weight. Participants who weigh more than or equal to 50 kilograms were administered every week, who weigh between 30 to less than 50 kg were administered every 10 days and who weigh less than 30 kg were administered every 2 weeks.
  Interventions: Combination Product: Belimumab

INTERVENTIONS:
Combination Product: Belimumab — Belimumab 200 mg/mL will be administered as SC injection in left or right thigh and the abdomen.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and pharmacodynamics (PD) of repeat doses of 200 milligrams per milliliter (mg/mL) belimumab administered via SC injection in pediatric participants 5 to 17 years of age with SLE on a background of standard of care therapy. This bridging PK study is part of an extrapolation strategy to support the use of SC belimumab in pediatric SLE participants, based on the completed adult SLE study with SC belimumab and the pediatric SLE study with intravenous (IV) belimumab. Part A is an open label 12-week treatment phase where participants will be enrolled and allocated to treatment cohorts based on their body weight at baseline. The dose and dosing regimens selected for SC administration in this pediatric population are intended to achieve a similar average exposure as observed with the weekly 200 mg SC dosing regimen in adult SLE patients. Part B is an optional 40-week open-label continuation phase, open to all participants who have completed Part A. Dosing of SC belimumab may continue at the same frequency in Part B or may require a change in frequency according to changes in participant body weight. The total duration of the study will be 68 weeks including a 12-Week open label treatment phase (Part A), an optional 40-week open-label continuation phase (Part B) and 16-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between 5 and 17 years of age inclusive, at the time of Day 1.
* Participants who meet the 1997 American College of Rheumatology (ACR) criteria for the classification of SLE;

  * Have or have had in series 4 or more of the 11 ACR criteria for the classification of SLE.
* Have active SLE disease defined as a safety of estrogen in lupus erythematosus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) score >=6 at screening.
* Have documented positive autoantibody test results within the study screening period, defined as an anti-nuclear antibody (ANA) titre >= 1:80 and/or a positive anti-dsDNA (>=30 international units per milliliter [IU/mL]) serum antibody test based on either the study's central laboratory results or the local laboratory results. Only unequivocally positive values as defined in the laboratory's reference range are acceptable; borderline values will not be accepted
* Are on a stable SLE treatment regimen, "Stable treatment at Baseline" consists of any of the following medications (alone or in combination) administered for a period of at least 30 days prior to Day 1;

  * Corticosteroids [prednisone or prednisone equivalent up to 0.5 milligram per kilogram per day (mg/kg/day)], for those participants on alternating day doses of steroids, use the average of 2 daily doses to calculate the average daily steroid dose.
  * Other immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium), calcineurin inhibitors (e.g. tacrolimus, cyclosporine), sirolimus, oral cyclophosphamide, 6-mercaptopurine or thalidomide.
  * Anti-malarials (e.g. hydroxychloroquine, chloroquine, quinacrine).
  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * New SLE therapy must not be added within 30 days of Day 1.
* Body weight >=15 kg.
* Male and/or female;

  * Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
  * No contraceptive measures are required for male participants.
  * A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies, Is not a woman of childbearing potential (WOCBP) or Is a WOCBP and is using a contraceptive method that is highly effective, with a failure rate of <1%, during the belimumab treatment period and for at least 16 weeks, corresponding to the time needed to eliminate any study intervention(s) (e.g., 5 terminal half-lives), after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
  * A WOCBP must have a negative highly sensitive pregnancy test (serum or as required by local regulations) within 35 days before the first dose of belimumab.
  * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Participant signs and dates a written age appropriate assent form (in accordance with applicable regulations) and the parent or legal guardian (or emancipated minor) that has the ability to understand the requirements of the study, provides written informed consent (including consent for the use and disclosure of research-related health information) that the participant will comply with the study protocol procedures (including required study visits).

Exclusion Criteria:

* Have an estimated glomerular filtration rate (eGFR) as calculated by Schwartz Formula of less than 30 milliliter/minute (mL/min).
* Have acute severe nephritis defined as significant renal disease (e.g., the presence of urinary sediments and other laboratory abnormalities) that, in the opinion of the study investigator, may lead to the participant requiring induction therapy during the first 12 weeks of the trial.
* Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoetic stem cell/marrow transplant.
* Have clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the participant at undue risk.
* Have a planned surgical procedure or a history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the participant unsuitable for the study.
* Have a history of malignant neoplasm within the last 5 years.
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months, or who in the investigator's opinion, pose a significant suicide risk.
* Have a history of a primary immunodeficiency.
* Have an immunoglobulin A (IgA) deficiency (IgA level <10 milligrams per deciliter [mg/dL]).
* Have acute or chronic infections requiring management, as follows;

  * Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
  * Use of parenteral [IV or Intramuscular (IM)] antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) for infection within 60 days of Day 1.
* Have a Grade 3 or greater laboratory abnormality based on the protocol defined adverse event and laboratory value severity grade scale except for the following that are allowed;

  * Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
  * Stable Grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy.
  * Stable Grade 3 hypoalbuminemia due to lupus nephritis, and not related to liver disease or malnutrition.
  * Any grade proteinuria.
  * Stable Grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis, and not related to alcoholic liver disease, uncontrolled diabetes or viral hepatitis. If present, any abnormalities in the alanine amininotransferase (ALT) and or aspartate aminotransferase (AST) must be <= Grade 2.
  * Stable Grade 3 neutropenia; or stable Grade 3 lymphopenia; or stable Grade 3 leukopenia, due to SLE.
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Have ever received treatment with belimumab.
* Have received any of the following within 364 days of Day 1;

  * Treatment with any B-cell targeted therapy [e.g., rituximab, other anti-CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], B lymphocyte stimulator (BLyS)-receptor fusion protein [BR3], transmembrane activator attached to the Fc portion of an immunoglobulin [TACI Fc]).
  * Abatacept.
  * Any biologic investigational agent.
* Have required 3 or more courses of systemic corticosteroids for concomitant conditions (e.g., asthma, atopic dermatitis) within 90 days of Day 1 (topical or inhaled steroids are permitted).
* Have received any of the following within 90 days of Day 1;

  * Anti-tumor necrosis factor (TNF) therapy (e.g., adalimumab, etanercept, infliximab).
  * Interleukin-1 receptor antagonist (anakinra).
  * Intravenous immunoglobulin (IVIG).
  * Plasmapheresis.
* Have received any of the following within 30 days of Day 1;

  * IV cyclophosphamide.
  * A non-biologic investigational agent (30 day window or 5 half-lives, whichever is greater).
  * Any new immunosuppressive/immunomodulatory agent.
  * High dose prednisone or equivalent (>1.5 mg/kg/day) or any intramuscular or intravenous steroid injection.
* Have received a live or live-attenuated vaccine within 30 days of Day 1.
* Have active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis or CNS vasculitis) requiring therapeutic intervention within 60 days of Day 1.
* Have required renal replacement therapy (e.g. hemodialysis, peritoneal dialysis) within 90 days of Day 1 or are currently on renal replacement therapy.
* Participation in an interventional clinical study either concurrently or within 6 months of screening. Participation in an observational study may be permitted.
* Positive immunodeficiency virus (HIV) antibody test
* Hepatitis B: Serologic evidence of Hepatitis B (HB) infection defined as Hepatitis B surface antigen positive (HBsAg+) or Hepatitis B core antibody positive (HBcAb+)
* Hepatitis C: Positive test for Hepatitis C antibody confirmed on an additional blood sample by ribonucleic acid (RNA) polymerase chain reaction (PCR) assay. Participants who are positive for Hepatitis C antibody and negative when the Hepatitis C RNA-PCR assay is performed on an additional sample will be eligible to participate. Participants who are positive for Hepatitis C antibody and have a positive result for the Hepatitis C virus (HCV) when the Hepatitis C RNA PCR assay is performed on the additional sample will not be eligible to participate. (Institution or country specific guidelines for blood sample volume limits must be followed in collection of the additional blood sample).
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 1.
* Are unable or unlikely, in the opinion of the investigator, to administer belimumab by SC injection and have no reliable source to administer the injection
* Children in Care: A Child in Care (CiC) is a child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The determination of whether a child meets the definition of CiC should be made with the study centre staff in consultation with the responsible institutional review board (IRB)/Ethics Committee.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2027-04-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- GSK Investigational Site, Cincinnati, Ohio, United States
- GSK Investigational Site, Rosario, Argentina
- Germany (2):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Saint Augustin
- Japan (2):
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
- GSK Investigational Site, San Luis Potosí City, Mexico
- GSK Investigational Site, Rotterdam, Netherlands
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Brunner HI, Anton J, Calvo-Penades I, Dimelow R, Horneff G, Kamphuis S, Marino R, van Maurik A, Minden K, Mori M, Ocran-Appiah J, Wilkinson C, Yamasaki Y, Assudani D; Pediatric Rheumatology Collaborative Study Group (PRCSG) and Paediatric Rheumatology International Trials Organisation (PRINTO) Network investigators. Pharmacokinetics, Pharmacodynamics, and Safety of Subcutaneous Belimumab in Pediatric Patients With Systemic Lupus Erythematosus: A Multicenter, Open-Label Trial. Arthritis Care Res (Hoboken). 2025 Nov 19. doi: 10.1002/acr.25700. Online ahead of print. PMID 41261055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 participants were screened and 25 were enrolled to the study. The primary study included Part A which is an open label 12-week treatment phase and Part B an optional 40-week open-label continuation phase, open to all participants who have completed Part A. An optional access extension phase is ongoing.
Pre-assignment Details: The data collection for the access extension phase is still ongoing and additional data will be provided after study completion date is achieved.
Period: Part A (Up to Week 12)
Arm/Group | Belimumab 200 mg
Started | 25
Completed | 25
Not Completed | 0
Period: Part B (Up to Week 52)
Arm/Group | Belimumab 200 mg
Started | 25
Completed | 23
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — INVESTIGATOR DISCRETION | 1
Period: Access Extension Phase
Arm/Group | Belimumab 200 mg
Started | 11 (Participants who completed Part B and entered access extension phase.)
Completed | 0
Not Completed | 11
Not completed — Ongoing | 11

BASELINE CHARACTERISTICS:
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 14.0 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 3
  ASIAN | 4
  BLACK OR AFRICAN AMERICAN | 1
  WHITE | 16
  MIXED RACE | 1

OUTCOME MEASURES:

1. Primary Outcome: Observed Belimumab Concentrations at Week 12
Description: Blood samples were collected for measurement of serum concentrations of belimumab. Observed belimumab concentrations at Week 12 is presented.
Time Frame: At Week 12
Population: The analysis was performed on the pharmacokinetic (PK) set that included all participants assigned treatment who received at least one dose of study treatment and for whom at least one post belimumab treatment PK sample was obtained and analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (ug/ml)
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
microgram per milliliter (ug/ml) | 106.42 [87.80 to 128.99]

2. Primary Outcome: Estimated Average Concentration (Cavg) of Belimumab at Steady State
Description: Blood samples were collected for measurement of serum concentrations of belimumab at steady state. Average concentrations were analyzed and reported for all time-points from Week 1 through Week 60.
Time Frame: Pre dose on Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52, and Week 60
Population: The analysis was performed on the PK Set that included all participants assigned treatment who received at least one dose of study treatment and for whom at least one post belimumab treatment PK sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
ug/ml | 124 (37.3)

3. Primary Outcome: Estimated Maximum Concentration (Cmax) of Belimumab at Steady State
Description: Blood samples were collected for measurement of serum concentrations of belimumab at steady state. Cmax was analyzed and reported for all time-points from Week 1 through Week 60.
Time Frame: Pre dose on Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52, and Week 60
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
ug/ml | 131 (34.9)

4. Primary Outcome: Estimated Minimum Concentration (Cmin) of Belimumab at Steady State
Description: Blood samples were collected for measurement of serum concentrations of belimumab at steady state. Cmin was analyzed and reported for all time-points from Week 1 through Week 60.
Time Frame: Pre dose on Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 52, and Week 60
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
ug/ml | 112 (41.7)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 68
Population: The safety analysis was performed on the Intent-To-Treat (ITT) set that included all participants assigned treatment who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
Participants | 22

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death.
Time Frame: Up to Week 68
Population: The safety analysis was performed on the ITT set that included all participants assigned treatment who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
Participants | 1

7. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESI included post-injection systemic reactions and hypersensitivity reactions, infections, malignancies, and depression/suicidality/self-injury. AESIs were followed until the event is resolved, stabilized, otherwise explained, or the participant is lost to follow-up.
Time Frame: Up to Week 68
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
Participants
  Malignancies | 0
  Post-Injection Systemic Reactions | 3
  Infections | 0
  Depression/Suicide/Self-injury | 0

8. Secondary Outcome: Percent Change From Baseline in Complement C3 and Complement C4 at Week 12 and Week 52
Description: Blood samples were collected from participants to assess complement C3 and complement C4 levels. Baseline status are defined as low complement [C3 less than (<) 90 milligrams per deciliter (mg/dL)] or normal/high (C3 >= 90 mg/dL) and low (C4 < 13 mg/dL) or normal/high (C4 >= 13 mg/dL) respectively. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 and 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: The analysis was performed on the ITT set that included all participants assigned treatment who received at least one dose of study treatment. Participants who had low baseline C3 and C4 levels were included in the respective analysis. Number of participants analyzed signifies those participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 15
Percent change
  Complement C3 (Week 12): number analyzed (Participants) | 11
  Complement C3 (Week 12) | 8.26 [2.0 to 24.8]
  Complement C3 (Week 52): number analyzed (Participants) | 11
  Complement C3 (Week 52) | 23.46 [-7.6 to 61.6]
  Complement C4 (Week 12) | 31.03 [-3.5 to 67.3]
  Complement C4 (Week 52): number analyzed (Participants) | 14
  Complement C4 (Week 52) | 67.52 [21.8 to 443.2]

9. Secondary Outcome: Percent Change From Baseline in Anti-Double Stranded Deoxyribonucleic Acid (dsDNA) Antibodies at Week 12 and Week 52
Description: Blood samples were collected for anti-dsDNA- antibody biomarker analysis. Baseline status are defined as positive (Anti-dsDNA antibody >= 30 International Units Per Milliliter (IU/mL)) or negative (Anti-dsDNA antibody< 30 IU/mL). Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 and 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: The analysis was performed on the ITT set that included all participants assigned treatment who received at least one dose of study treatment. Participants who had positive anti-dsDNA antibody levels at baseline were included in the analysis. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 15
Percent change
  Week 12 | -17.74 [-68.0 to 40.0]
  Week 52: number analyzed (Participants) | 14
  Week 52 | -58.88 [-85.3 to -2.4]

10. Secondary Outcome: Percent Change From Baseline in CD19+ Total B Cells and CD20+ B Cells at Week 12 and Week 52
Description: Blood samples were collected for biomarker analysis. B cell subsets included CD19+ total B cells and CD 20+ B cells. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 and 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: The analysis was performed on the ITT set that included all participants assigned treatment who received at least one dose of study treatment. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 15
Percent change
  CD19+ Total B cells (Week 12) | -42.97 [-74.4 to 68.8]
  CD19+ Total B cells (Week 52): number analyzed (Participants) | 14
  CD19+ Total B cells (Week 52) | -61.32 [-89.4 to 95.5]
  CD20+ B cells (Week 12) | -41.85 [-75.8 to 92.1]
  CD20+ B cells (Week 52): number analyzed (Participants) | 14
  CD20+ B cells (Week 52) | -61.65 [-89.9 to 92.3]

11. Secondary Outcome: Percent Change From Baseline in Naïve B Cells and Memory B Cells at Week 12 and Week 52
Description: Blood samples were collected for biomarker analysis and included CD20+ CD27- Naïve B cells and CD20+ CD27+ memory B cell. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 and 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 15
Percent change
  Naïve B Cells (Week 12) | -53.19 [-81.5 to 21.0]
  Naïve B Cells (Week 52): number analyzed (Participants) | 14
  Naïve B Cells (Week 52) | -72.13 [-94.5 to 20.3]
  Memory B Cells (Week 12) | 69.06 [-36.7 to 531.8]
  Memory B Cells (Week 52): number analyzed (Participants) | 14
  Memory B Cells (Week 52) | 27.10 [-63.2 to 402.9]

12. Secondary Outcome: Percent Change From Baseline in in CD27bright CD38bright Plasma Blasts at Week 12 and Week 52
Description: Blood samples were collected for CD27bright CD38bright Plasma blasts biomarker analysis. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 and 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 15
Percent change
  Week 12 | 9.40 [-81.8 to 428.1]
  Week 52: number analyzed (Participants) | 14
  Week 52 | -70.07 [-88.9 to 193.1]

13. Secondary Outcome: Percent Change From Baseline in Immunoglobulin A (IgA), Immunoglobulin G (IgG) and Immunoglobulin M (IgM) at Week 12
Description: Blood samples were collected for analysis of immunoglobulins: Immunoglobulin A (IgA), Immunoglobulin G (IgG), and Immunoglobulin M (IgM). Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 12 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 25
Percent change
  Immunoglobulin A (IgA) | -3.13 [-35.2 to 8.0]
  Immunoglobulin G (IgG) | -3.40 [-30.7 to 12.7]
  Immunoglobulin M (IgM) | -10.41 [-49.2 to 4.3]

14. Secondary Outcome: Percent Change From Baseline in Immunoglobulin A (IgA), Immunoglobulin G (IgG) and Immunoglobulin M (IgM) at Week 52
Description: Blood samples were collected for analysis of immunoglobulins: Immunoglobulin A (IgA), Immunoglobulin A (IgG), and Immunoglobulin M (IgM). Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline value X 100.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 200 mg
Number analyzed (Participants) | 21
Percent change
  Immunoglobulin A (IgA) | -13.06 [-37.5 to 41.0]
  Immunoglobulin G (IgG) | -12.29 [-34.0 to 10.6]
  Immunoglobulin M (IgM) | -30.79 [-56.7 to -8.9]

ADVERSE EVENTS:
Time Frame: Up to Week 68 (treatment: up to 52 weeks [12 weeks Part A; 40 weeks Part B extension phase] and follow-up: 16 weeks)
Description: The safety analysis was based on the Intent-To-Treat set that comprised of all participants assigned treatment who received at least one dose of study treatment.
Arm/Group | Belimumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 200 mg (N=25)
COVID-19 (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 200 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Injection site erythema (General disorders) | 2 (3)
Injection site pain (General disorders) | 4 (9)
COVID-19 (Infections and infestations) | 8 (8)
Nasopharyngitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Urine protein/creatinine ratio increased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04179032/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT04179032/SAP_001.pdf